CLINICAL TRIAL: NCT07080567
Title: Maraviroc for Stroke Recovery (MASTER): A Phase 2 Double-Blind Placebo-Controlled Randomized Clinical Trial
Brief Title: Manipulating the Peri-Infarct Area Using Maraviroc to Enhance Motor Skills After Stroke
Acronym: MASTER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emmanuel Carrera (Other)
Responsible Party: Sponsor-Investigator, Emmanuel Carrera, Sponsor-Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-02359; 215285 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2025-07-02; First posted 2025-07-23 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke; Stroke; Stroke Acute
Keywords: Ischemic Stroke; Maraviroc; CCR5; Stroke; Stroke Acute; Motor Recovery; Randomized Controlled Trial
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Maraviroc; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maraviroc (Active Comparator): Maraviroc (Celsentri) 300 mg twice daily
  Interventions: Drug: Maraviroc
- Placebo (Placebo Comparator): Placebo (Mannitol) encapsulated
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Maraviroc — Maraviroc (300mg) twice daily for 90 days
  Other Names: Celsentri
  Arms: Maraviroc
Drug: Mannitol — Placebo intervention
  Arms: Placebo

SUMMARY:
MASTER is a single-center, patient and investigator-blinded, Randomized Controlled Trial (RCT) to compare the efficacy of Maraviroc, a C-C chemokine receptor 5 (CCR5) antagonist, against placebo regarding motor function and motor learning skills in the first 3 months after ischemic stroke.

DETAILED DESCRIPTION:
Stroke is a common disease and one of the leading causes of death and disability worldwide. Despite advances in acute stroke therapies (intravenous thrombolysis and/or mechanical thrombectomy), deficits remain frequent after stroke. Pharmacological approaches have the benefit of being independent of patient participation, are easily administered, and involve limited medical resources. Unfortunately, the efficacy of several drugs that improve behavioural in preclinical models have yet to be confirmed in humans. Maraviroc, a C-C chemokine receptor 5 (CCR5) antagonist has shown promise in preclinical models, and instead of targeting neurotransmitters, is believed to augment rehabilitation by decreasing infarct size, increasing neuroplasticity, and most importantly, improving behaviour.

The MASTER trial is a single-center, double-blinded, randomized placebo-controlled, phase II clinical trial designed to evaluate the efficacy of Maraviroc (Celsentri) compared to a placebo, in improving outcomes following ischemic stroke in the early stage of recovery. 80 patients will be recruited within 5 days of stroke onset, and will receive either Maraviroc or a placebo drug for 90 days.

Participants will be assessed using a combination of clinical measurements, motor tests, and biometrics throughout the 90 days of intervention, and upon follow-up at 6-months post stroke onset. Several types of brain images will be obtained before and after the intervention period (day 0 and day 90), and participants will also perform a motor learning task before and after the intervention period (day 0 and day 90). Study personnel and participants will be blinded to the treatment, which will be randomly assigned to an intervention group with stratification based on side of the infarct and motor deficit.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* ≥18 years at time of signing of informed consent
* Acute ischemic stroke.
* Stroke onset < 7 days from randomization.
* Contralateral, unilateral, incomplete upper limb paresis, incl. :
* FMA-UE < 63/66
* Residual voluntary finger extension (VFE) of > 10 degrees

Exclusion Criteria:

* Pregnancy/lactation or positive pregnancy test in women of childbearing age
* Pre-stroke handicap (mRS > 2)
* Diseases affecting motor function (e.g., Parkinson's Disease, Amyotrophic Lateral Sclerosis (ALS))
* Participation in another study with investigational medicinal product within 30 days preceding and during the present study
* Enrolment of the investigator, his/her family members, employees, or other dependent persons
* Known hypersensitivity to Maraviroc, Mannitol, peanuts, or soy
* History of significant liver disease, hepatitis, elevated liver function tests (> 1.5 upper limit of normal)
* History of significant renal disease or End Stage Renal Disease/dialysis, acute renal injury, Creatinine Clearance (CrCl < 30ml/min/1.73m2)
* Patients with cardiovascular comorbidities and risk for orthostatic hypotension
* HIV infection
* Concomitant use of strong CYP3A4 inhibitors or inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Upper Extremity Fugl-Meyer Assessment (FMA-UE) Score | Day 90
  Reliable and validated score of motor function of the upper extremities after stroke. Range: 0-66, higher values indicating better motor function.

SECONDARY OUTCOMES:
Motor Learning Score | Day 0, 90
  A motor sequence learning score assessing the capability of the participant to learn a finger tapping sequence of 6 items.
Number of adverse events (AE) of special interest | Day 0-180 (inclusive)
  The number of patients experiencing AE of special interest : MACE (Major Adverse Cardiovascular Events) - Acute myocardial infarction ; Acute coronary syndrome ; Stroke ; Heart failure ; All cause death ; Cardiovascular death ; Revascularization AND any liver adverse events AND any infection adverse events. Assesed by: CTCAE v5.0
Number of Serious Adverse Events (SAE) | 0-180 days (inclusive)
  Number of any SAEs occuring during the study follow-up. Assessed by: CTCAE v5.0.

OTHER OUTCOMES:
9-hole Peg Test (Time) | Day 0, 30, 60, 90, and 180.
  The 9-hole peg test is used to measure dexterity. It is measured in seconds to complete the task, with lower duration indicating better dexterity.
Pinch force | Day 0, 30, 60, 90, and 180.
  Pinch force will be measured using a finger dynamometer, measured in kg. A greater value indicates greater finger strength.
Grip strength | Day 0, 30, 60, 90, and 180.
  Grip strength will be measured using a hand dynamometer. Strength is measured in kg, with a greater value indicating stronger grip strength.
National Institute of Health Stroke Scale (NIHSS) | Day 0, 30, 60, 90, 180
  A 15-item neurologic examination stroke scale (0 - 42), with higher scores indicating greater neurological impairment.
Modified Rankin Scale (mRS) | Day 0, 30, 60, 90, 180
  An ordinal scale measuring degree of dependence and disability following stroke, ranging from 0 to 6. A lower score indicates greater independence and less disability. 6 indicates death.
Barthel Index | Day 0, 30, 60, 90, 180
  A scale measuring independence for activities of daily living, on a scale from 0 to 100. Higher scores indicate greater functional independence.
Functional brain connectivity | Day 0, 90
  Correlated Blood Oxygen Level Dependent (BOLD) imaging responses in the brain derived from resting state functional MRI scanning (values from 0 to 1, greater values indicating more connectivity), focussing on core motor and peri-infarct functional connectivity.
Structural brain connectivity | Day 0, 90
  Diffusion weighted imaging (DWI) derived structural connectivity, measured as fractional anisotropy of connecting tracts (values of 0 to 1, higher values indicating more directed water diffusion) , focussing on core motor and peri-infarct connectivity.
Neurite Density Index | Day 0, 90
  Microstructure analysis of the brain derived from a multi-shell Diffusion Weighted Imaging (DWI) MRI sequence, using a neurite density index (0 - 1). Greater values indicate greater density of neurites.
Brain metabolite concentrations | Day 0, 90
  Measurement of brain metabolite concentrations - N-acetylaspartate (NAA), Glutamate-Glutamine complex (Glx), Gamma-aminobutyric Acid (GABA), Creatinin (Cr) - using whole-brain magnetic resonance spectroscopic imaging (MRSI).

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Carrera, MD, Principal Investigator — Hôpitaux Universitaires Genève
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized patient data of the primary and secondary study outcomes (FMA-UE, global functioning scores, motor learning scores) are currently anticipated to be shared dependent on participant consent to data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The IPD and supporting information will be available following the publication of the results (est. 2028) and will be available indefinitely.
Access Criteria: IPD will be available in a de-identified format to ensure participant confidentiality. Access will be granted to qualified researchers upon reasonable request, subject to prior approval by the sponsor and the demonstration of approval from a competent ethics committee. The shared data will include de-identified IPD that underlies the results reported in the publication (text, tables, figures, and appendices). Supporting documents such as the study protocol, statistical analysis plan, and clinical study report may also be available. Data will be accessible through a secure platform or via direct request after publication of the main study results.

REFERENCES:
- [Background] Joy MT, Ben Assayag E, Shabashov-Stone D, Liraz-Zaltsman S, Mazzitelli J, Arenas M, Abduljawad N, Kliper E, Korczyn AD, Thareja NS, Kesner EL, Zhou M, Huang S, Silva TK, Katz N, Bornstein NM, Silva AJ, Shohami E, Carmichael ST. CCR5 Is a Therapeutic Target for Recovery after Stroke and Traumatic Brain Injury. Cell. 2019 Feb 21;176(5):1143-1157.e13. doi: 10.1016/j.cell.2019.01.044. PMID 30794775
- [Background] Sharif A, Jeffers MS, Fergusson DA, Bapuji R, Nicholls SG, Humphrey J, Johnston W, Mitchell E, Speirs MA, Stronghill L, Vuckovic M, Wulf S, Shorr R, Dowlatshahi D, Corbett D, Lalu MM. Preclinical systematic review of CCR5 antagonists as cerebroprotective and stroke recovery enhancing agents. Elife. 2025 Apr 7;14:RP103245. doi: 10.7554/eLife.103245. PMID 40193175